CLINICAL TRIAL: NCT01676311
Title: Huperzine A for the Treatment of Cognitive, Mood, and Functional Deficits After Moderate and Severe TBI
Brief Title: Effects of Huperzine A in Treatment of Moderate to Severe TBI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual rate: 14 participants enrolled (target of 30).
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Ross D. Zafonte, MD, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-p-002490
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Traumatic Brain Injury
Keywords: cognition; seizures; electroencephalography; transcranial magnetic stimulation; huperzine; chinese club moss
MeSH Terms: conditions — Brain Injuries, Traumatic; Seizures | interventions — huperzine A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Huperzine A (Experimental): Huperzine A will be administered to patients, titrating dose up from 100mcg/day to 600mcg per day over the course of 20 days - and remaining on the dose of 600mcg/day for the remainder of the drug phase (64 days) - for a total of 12 weeks on Huperzine A.
  Interventions: Drug: Huperzine A
- Placebo (Placebo Comparator): Placebo will be administered to patients at the same frequency/intervals as the experimental arm (Huperzine-A).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Huperzine A — Huperzine A will be administered for 12 weeks as outlined in the Arm Description
  Other Names: huperzia serrata; chinese club moss
  Arms: Huperzine A
Drug: Placebo — Placebo Arm (blinded randomization) for Huperzine A Intervention
  Arms: Placebo

SUMMARY:
We will explore the use of Huperzine A in patients who have sustained a moderate to severe Traumatic Brain Injury. We aim to determine whether Huperzine A, as compared with placebo, would have an effect on memory function after TBI. Additionally, we aim to determine whether use of Huperzine A in these patients can change brain activity (as indexed by EEG and Transcranial Magnetic Stimulation - TMS), and reduce prevalence/frequency of post-traumatic seizures. We also aim to evaluate the safety of Huperzine A in this population as compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 65
* Moderate or severe TBI, based on admission Emergency Room GCS 3-12
* All subjects will be greater than 2 weeks, but no more than 1 year, after the qualifying TBI, and will be symptomatic at enrollment (i.e. all subjects will exhibit evidence of ongoing posttraumatic amnesia via the Galveston Orientation Amnesia test (GOAT), or score at least 1.5 SD below the mean for completion time on Part B of the Trail Making Test.
* Agreement to undergo no changes in concomitant medications (including dietary supplements) or therapeutic interventions during the first 12 weeks of the study (that is, the 12 weeks of dosing with study drug), except where medically indicated. Stable concomitant drug regimen (greater than two weeks pre-enrollment without changes)
* Normal swallowing
* English-speaking (since not all of the outcome metrics are normed outside of the English language)
* Patient can be on seizure medication.

Exclusion Criteria:

* Patients taking acetylcholinesterase inhibitors and other cholinergic and anticholinergic drugs (e.g., tacrine, physostigmine, velnacrine, donepezil, rivastigmine, metrifonate) and CYP1A inducing drugs.
* Evidence of more than 1 seizure in the past 4 weeks prior to enrollment: Patients may not be enrolled if there is evidence of more than one seizure (clinical or electrographic, but not including epileptiform or other irritative discharges) during the 4 weeks prior to enrollment.
* Premorbid history of epilepsy with seizure frequency >1 per month: Patients with a history of idiopathic epilepsy may not be enrolled if their seizure frequency was > 1 per month in the 3 months prior to injury. If pre-injury seizure frequency was < 1 per month but there is documented evidence that post-injury seizure frequency is > 1 per month or there is documented evidence of an increase in the severity or duration of a single seizure relative to the premorbid history, the patient must be excluded.
* Evidence of premorbid major CNS disorder, developmental disorder, psychiatric disorder or substance abuse: Prior to sustaining TBI, patient was diagnosed and/or treated for a major neurologic condition, pervasive developmental disorder (e.g., mental retardation, autism), psychiatric disorder or substance abuse that continued to produce functional disability up to the time of injury.
* Individuals with disorders of consciousness, as defined at the time of screening of having vegetative and/or minimally conscious state, will not be enrolled. However, these patients may be followed until they:

  * Meet eligibility criteria
  * Are more than 12 weeks post injury
  * Are discharged
* Pregnancy, as determined by urine hCG testing before randomization
* Breast feeding females
* Significant hematologic, renal or hepatic dysfunction [Hepatic/renal dysfunction is generally identified as lab results > two times the upper limits of normal (ULN), and hematologic dysfunction is determined by clinically significant abnormal lab results], on baseline laboratory examination.
* Slow heart rate (bradycardia) or other heart conditions related to rate
* History of peptic ulcer disease
* History of asthma or emphysema
* History of GI/urinary tract blockages (i.e. ileus, IBS)
* History of glaucoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Zafonte, DO, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Huperzine A | Placebo
Started | 7 | 7
Completed | 7 | 5
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Huperzine A | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.00 (16.21) | 38.57 (16.60) | 37.79 (15.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
Admission status [Count of Participants; unit: Participants]
  Inpatient | 1 | 4 | 5
  Outpatient | 6 | 3 | 9
Days post-injury [Mean (Standard Deviation); unit: days] | 155.40 (130.27) | 226.86 (120.30) | 197.08 (124.17)

OUTCOME MEASURES:

1. Primary Outcome: California Verbal Learning Test- 2nd Edition (CVLT-II): Learning and Memory
Description: Measure of learning and memory function. Three indices of the CVLT-II were calculated. The full name, abbreviated name, and the minimum and maximum possible scores of each index are indicated below:
  1. California Verbal Learning Test- 2nd Edition- Total Learning [CVLT-II-TL] (Minimum score=0; Maximum score= 80)
  2. California Verbal Learning Test- 2nd Edition- Short delay free recall [CVLT-II-SDFR] (Minimum score=0; Maximum score=16)
  3. California Verbal Learning Test- 2nd Edition- Long delay free recall [CVLT-II-LDFR] (Minimum score=0; Maximum score=16)
  High scores are indicative of greater memory and learning for each index (i.e. better outcome).
Time Frame: Baseline, 6 weeks, 12 weeks, 24 weeks and at 52 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Huperzine A | Placebo
Number analyzed (Participants) | 7 | 5
score on a scale
  CVLT-II-TL - Baseline | 28.57 (12.35) | 34.40 (18.73)
  CVLT-II-TL - Week 6 | 31.43 (11.37) | 45.00 (17.65)
  CVLT-II-TL - Week 12 | 38.29 (14.20) | 49.60 (18.27)
  CVLT-II-TL - Week 24 | 33.29 (14.29) | 44.60 (14.12)
  CVLT-II-TL - Week 52 | 37.43 (11.30) | 49.40 (15.00)
  CVLT-II-SDFR - Baseline | 3.86 (4.38) | 5.80 (4.66)
  CVLT-II-SDFR - Week 6 | 4.14 (3.53) | 7.83 (4.12)
  CVLT-II-SDFR - Week 12 | 6.29 (4.99) | 10.40 (5.46)
  CVLT-II-SDFR - Week 24 | 4.86 (4.45) | 10.00 (4.24)
  CVLT-II-SDFR - Week 52 | 5.43 (3.36) | 9.80 (5.50)
  CVLT-II-LDFR - Baseline | 5.00 (4.80) | 7.00 (5.70)
  CVLT-II-LDFR - Week 6 | 4.43 (4.39) | 8.33 (4.08)
  CVLT-II-LDFR - Week 12 | 6.00 (4.76) | 10.00 (5.96)
  CVLT-II-LDFR - Week 24 | 4.29 (4.46) | 8.40 (4.67)
  CVLT-II-LDFR - Week 52 | 6.14 (4.67) | 10.00 (4.74)
Statistical Analysis 1: Comparison: Huperzine A vs Placebo; Regression analysis was run incorporating group, CVLT-II-total learning score at baseline and week 12, and covariates (Beck Depression Index [BDI], time post-injury, British Columbia Postconcussion Symptom Inventory [BC-PSI]). Regression analyses were repeated, permuting data observations for each outcome. The BDI and BC-PSI are covariates in the regression model and not pre-specified Primary and Secondary Outcome Measures; Test type: Superiority; p = 0.38, Regression, Linear — For each permutation of the data, relevant result was saved and the corresponding p-value represents the proportion of results at least as extreme as observed in the original data
Statistical Analysis 2: Comparison: Huperzine A vs Placebo; Regression analysis was run incorporating group (Huperzine A, placebo), baseline CVLT-II-short delay free recall (SDFR) score, outcome (CVLT-II-SDFR at week 12) and covariates (Beck Depression Index, time post-injury, British Columbia Postconcussion Symptom Inventory). Regression analyses were repeated, permuting data observations for each outcome i.e. we permuted the labels (Huperzine A or placebo) among the data observations and re-ran the regression; Test type: Superiority; p = 0.38, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Huperzine A vs Placebo; Regression analysis was run incorporating group (Huperzine A, placebo), baseline CVLT-II-long delay free recall (LDFR) score, outcome (CVLT-II-LDFR at week 12) and covariates (Beck Depression Index, time post-injury, British Columbia Postconcussion Symptom Inventory). Regression analyses were repeated, permuting data observations for each outcome i.e. we permuted the labels (Huperzine A or placebo) among the data observations and re-ran the regression; Test type: Superiority; p = 0.42, Regression, Linear — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Amplitude of Event Related Potentials (ERPs) P50 and P300
Description: Event Related Potentials (ERPs): P50 and P300 are neurophysiological measurements that index cortical electrical activity associated with a given stimulus. P50 and P300 were measured using auditory stimuli. P50 represents an index of activity in the cholinergic system and has been used to characterize presynaptic cholinergic deficit. P300 is a measure of general cognitive processing elicited during attention, memory, and executive tasks.
Time Frame: Baseline, 12 Weeks
Population: Of the 12 participants who completed the 12-week treatment period, P50 and P500 amplitude data could be analyzed for 4 participants. Data for the other 8 participants could not be analyzed as the data were compromised by movement artifact during recording.
Measure: Median (Inter-Quartile Range); unit: mV
Arm/Group | Huperzine A | Placebo
Number analyzed (Participants) | 3 | 1
mV
  P300 Amplitude - Baseline | 13.57 [9.28 to 17.86] | 9.96
  P300 Amplitude - Week 12 | 12.69 [4.10 to 21.28] | 9.69
  P50 Amplitude - Baseline | 7.89 [4.59 to 11.19] | NA — The participant did not have P50 data that could be analyzed.
  P50 Amplitude - Week 12 | 5.89 [-0.36 to 12.14] | NA — The participant did not have P50 data that could be analyzed.

3. Secondary Outcome: Latency of Event Related Potentials (ERPs) P50 and P300
Description: Event Related Potentials (ERPs): P50 and P300 are neurophysiological measurements that index cortical electrical activity associated with a given stimulus. P50 and P300 were measured using auditory stimuli. P50 represents an index of activity in the cholinergic system and has been used to characterize presynaptic cholinergic deficit and P300 is a measure of general cognitive processing elicited during attention, memory, and executive tasks.
Time Frame: Baseline, 12 weeks
Population: Of the 12 participants who completed the 12-week treatment period, P50 and P500 latency data could be analyzed for 3 participants. Data for the other 9 participants could not be analyzed as the data were compromised by movement artifact during recording.
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Huperzine A | Placebo
Number analyzed (Participants) | 3 | 0
ms
  P300 Latency - Baseline | 309 [306 to 312] |
  P300 Latency - Week 12 | 311 [291 to 331] |
  P50 Latency - Baseline | 50 [48 to 52] |
  P50 Latency - Week 12 | 49 [49 to 49] |

4. Secondary Outcome: Number of Participants Who Experienced Post-traumatic Seizure During 12-week Treatment Window
Description: To determine whether Huperzine A changes the prevalence of post-traumatic seizure after moderate and severe TBI as compared to placebo at 12 weeks post-enrollment (immediate seizures prevalence).
Time Frame: Baseline and weekly for 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Huperzine A | Placebo
Number analyzed (Participants) | 7 | 5
Participants | 2 | 1
Statistical Analysis 1: Comparison: Huperzine A vs Placebo; Test type: Superiority; p = 0.48, Chi-squared test and permutation test — A chi-square test with factors of group (Huperzine A, placebo) and occurrence of seizure (yes, no) was performed. A permutation test was the used to assess the effect of Huperzine A on the prevalence of seizures

5. Secondary Outcome: Number of Participants With Self-reported Side Effects During 12-week Treatment Window
Description: To evaluate the safety and tolerability of Huperzine A in this patient population as compared to placebo the frequency of self-reported side effects during the 12-week treatment window were grouped categorically by system (behavioral, cardiac-respiratory, dermatological,gastrointestinal, genitourinary/neurological, hematological, musculoskeletal, neurological).
Time Frame: Baseline and weekly for 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Huperzine A | Placebo
Number analyzed (Participants) | 7 | 6
Participants
  Behavioral side effects | 5 | 4
  Cardiac-respiratory side effects | 6 | 4
  Dematological side effects | 2 | 0
  Gastrointestinal side effects | 3 | 1
  Genitourinary/neurological side effects | 1 | 1
  Hematological side effects | 6 | 6
  Musculoskeletal side effects | 3 | 2
  Neurological side effects | 7 | 5
Statistical Analysis 1: Comparison: Huperzine A vs Placebo; Behavioral side effects statistical analysis; Test type: Superiority; p = 0.44, Chi-squared test and permutation test — A chi-squared test with factors of group (Huperzine A, placebo) and occurrence of behavioral side effects (yes, no) were performed. A permutation test was used to assess the effect of Huperzine A on the incidence of behavioral side effects
Statistical Analysis 2: Comparison: Huperzine A vs Placebo; Cardiac-respiratory side effects statistical analysis; Test type: Superiority; p = 0.81, Chi-squared test and permutation test — A chi-squared test with factors of group (Huperzine A, placebo) and occurrence of cardiac-respiratory side effects (yes, no) were performed. A permutation test was used to assess the effect of Huperzine A on the incidence of these side effects
Statistical Analysis 3: Comparison: Huperzine A vs Placebo; Dermatological side effects statistical analysis; Test type: Superiority; p = 0.81, Chi-squared test and permutation test — A chi-squared test with factors of group (Huperzine A, placebo) and occurrence of dermatological side effects (yes, no) were performed. A permutation test was used to assess the effect of Huperzine A on the incidence of dermatological side effects
Statistical Analysis 4: Comparison: Huperzine A vs Placebo; Gastrointestinal side effects statistical analysis; Test type: Superiority; p = 0.73, Chi-squared test and permutation test — A chi-squared test with factors of group (Huperzine A, placebo) and occurrence of gastrointestinal side effects (yes, no) were performed. A permutation test was used to assess the effect of Huperzine A on the incidence of these side effects
Statistical Analysis 5: Comparison: Huperzine A vs Placebo; Genitourinary/neurological side effects statistical analysis; Test type: Superiority; p = 0.54, Chi-squared test and permutation test — A chi-squared test with factors of group (Huperzine A, placebo) and occurrence of genitourinary/neurological side effects (yes, no) were performed. A permutation test was used to assess the effect of Huperzine A on the incidence of these side effects
Statistical Analysis 6: Comparison: Huperzine A vs Placebo; Hematological side effects statistical analysis; Test type: Superiority; p = 0.27, Chi-squared test and permutation test — A chi-squared test with factors of group (Huperzine A, placebo) and occurrence of hematological side effects (yes, no) were performed. A permutation test was used to assess the effect of Huperzine A on the incidence of these side effects
Statistical Analysis 7: Comparison: Huperzine A vs Placebo; Musculoskeletal side effects statistical analysis; Test type: Superiority; p = 0.41, Chi-squared test and permutation test — A chi-squared test with factors of group (Huperzine A, placebo) and occurrence of musculoskeletal side effects (yes, no) were performed. A permutation test was used to assess the effect of Huperzine A on the incidence of these side effects
Statistical Analysis 8: Comparison: Huperzine A vs Placebo; Neurological side effects statistical analysis; Test type: Superiority; p = 1.00, Chi-squared test and permutation test — A chi-squared test with factors of group (Huperzine A, placebo) and occurrence of neurological side effects (yes, no) were performed. A permutation test was used to assess the effect of Huperzine A on the incidence of these side effects

ADVERSE EVENTS:
Time Frame: Telephone: Weekly from baseline to 12 weeks (active treatment phase). In-person follow-up visits: Baseline, 6, 12, 13, 24, and 52 weeks. Subjects were instructed to call the Study Coordinator if a serious adverse event occurred between scheduled telephone or in-person follow-ups.
Description: Adverse events were collected and recorded using a standard adverse event form that included 35 possible adverse events. For 'Adverse Events', 'Serious Adverse Events', and 'Other (Not Including Serious) Adverse Events', results are reported for all participants who were 'at risk' i.e. received Huperzine A or placebo and completed at least one telephone or in-person follow-up visit (Huperzine A group: 7 participants; Placebo group: 6 participants).
Arm/Group | Huperzine A | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Huperzine A (N=7) | Placebo (N=6)
Seizure (Nervous system disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Huperzine A (N=7) | Placebo (N=6)
Anxiety (Psychiatric disorders) | 4 | 4
Irritability (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 2 | 1
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased blood pressure (General disorders) | 6 | 4
Decrease in heart rate (General disorders) | 6 | 4
Skin rash (Skin and subcutaneous tissue disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Loss of appetite (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Increased saliva production (Gastrointestinal disorders) | 2 | 1
Incontinence (Renal and urinary disorders) | 1 | 1
Low white blood cell count (Blood and lymphatic system disorders) | 6 | 6
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1
Difficulty sleeping (General disorders) | 3 | 3
Confusion (Nervous system disorders) | 5 | 3
Headache (Nervous system disorders) | 3 | 2
Fatigue (General disorders) | 4 | 5
Thinking abnormalities (Nervous system disorders) | 2 | 2
Weakness (Nervous system disorders) | 1 | 2
Slurred speech (Nervous system disorders) | 0 | 2
Abnormal vision (Eye disorders) | 2 | 2
Light sensitivity (Nervous system disorders) | 1 | 1
Increased uncontrolled movement (Nervous system disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Enrollment - not able to enroll target N, therefore small number of subjects analyzed.

Neurophysiologic measures - difficulty collecting data from subjects for several reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT01676311/Prot_SAP_000.pdf